CLINICAL TRIAL: NCT05035134
Title: Application of Circulating Exosomes in Early Diagnosis and Prognosis Evaluation After Intracerebral Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDSJWKICHEX
Record Dates: First submitted 2021-07-26; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Intracerebral Hemorrhage；Circulating Exosomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to observe the relationship between the changes of circulating exosomes and the development and outcome of the disease in patients with intracerebral hemorrhage, and to search for early serum markers and potential intervention targets for disease monitoring in patients with intracerebral hemorrhage

ELIGIBILITY:
Inclusion Criteria:

1. No systematic treatment was given before admission;
2. The patients were diagnosed with cerebral hemorrhage, and had imaging evidence;
3. The age was more than 18 years old;
4. The patient or family member agrees to sign the informed consent.

Exclusion Criteria:

1. Hematoma is caused by secondary factors (intracranial tumor, arteriovenous malformation or aneurysm);
2. Bleeding into the ventricle;
3. Multiple cerebral hemorrhage;
4. The patient did not receive treatment in our hospital;
5. Severe disability, dementia, or organ dysfunction before onset
6. Coagulopathy or long-term use of anticoagulants
7. Hematoma affects brain stem
8. Subjects refused to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All of the ICH patients receiving treatment in Tangdu Hospital during 2021-2022
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-12 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
The type and content of circulating exosomes | within 24 hours of ICH
  After the exosomes were isolated, RNA sequencing and proteome sequencing were performed to identify the change of circulating exosomes
Modified Rankin scale (mRS) scores | from onset to three months or six months
  mRS scores was divided into seven grades (0-6). The higher the score, the more severe the symptoms

SECONDARY OUTCOMES:
mortality | through study completion，an average of 1 year
hospital stay | From hospitalization to discharge，up to one month

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qu, M.D, Ph.D, Study Chair — Tang-Du Hospital; Xun Wu, M.D, Principal Investigator — Tang-Du Hospital
Locations (1):
- Tandu Hospital, Fourth Military Medical University, Xi'an, China